CLINICAL TRIAL: NCT03388593
Title: A Multi-center, Randomized, Double-blined, Placebo Parallel Controlled Phase III Clinical Trial to Evaluate the Effect of Injectable Neucardin on the Mortality of Subjects With Chronic Systolic Heart Failure on Standard HF Therapy.
Brief Title: Survival Study of the Recombinant Human Neuregulin-1β in Subjects With Chronic Heart Failure.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-01-306
Record Dates: First submitted 2017-12-19; First posted 2018-01-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; neuregulin; mortality
MeSH Terms: conditions — Fibromatosis, Gingival, 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo in addition to standard therapy
  Interventions: Drug: Placebo
- rhNRG-1 (Experimental): rhNRG-1 in addition to standard therapy
  Interventions: Drug: rhNRG-1

INTERVENTIONS:
Drug: rhNRG-1 — 10 hours per day i.v drip for the first 10 days (0.6ug/kg/day), followed by weekly 10 minutes i.v bolus (0.8ug/kg/day), from the 3rd week for 23 weeks
  Other Names: Neucardin™
  Arms: rhNRG-1
Drug: Placebo — 10 hours per day i.v drip for the first 10 days (0ug/kg/day), followed by weekly 10 minutes i.v bolus (0ug/kg/day), from the 3rd week for 23 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy of rhNRG-1 in reducing the death rate of heart failure subjects with baseline NT-proBNP level between 600 pg/ml and 1700 pg/mL and NYHA class II to III.

DETAILED DESCRIPTION:
The mortality of chronic heart failure patients remains high, in spite of current treatment. RhNRG-1(recombinant human neuregulin-1)directly work on the cardiomyocyte and restored the normal structure and function of it. Both the preclinical trials, phase II clinical trials and already completed phase III clinical trails have confirmed that rhNRG-1 effectively enhance the heart function, reverse the remodeling of left ventricular, and reduce all-cause mortality in heart failure animals and humans. More importantly, rhNRG-1 can significantly reduce the mortality of heart failure subjects with baseline NT-proBNP level ≤1600 fmol/mL and NYHA class II to III. In this phase III study, the investigators will further confirm the efficacy of rhNRG-1 in reducing the death rate of heart failure subjects with baseline NT-proBNP level between 600 pg/ml and 1700 pg/mL and NYHA class II to III.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 75, gender balance (no more than 960 subjects of either gender in total 1600 subjects).
* 2. Left ventricular ejection fraction (LVEF)≤40% (ECHO).
* 3. Subjects with chronic heart failure (NYHA class II OR III ).
* 4. 600 pg/ml ≤NT-proBNP≤1700 pg/ml ( by Roche assay Kit in central lab).
* 5. Diagnosed as chronic systolic heart failure (history, symptoms, signs), and in stable condition in the last one month.
* 6. Receiving standard therapy for chronic heart failure, reach target dose or max tolerable dose for one month, or has not changed the dose for one month before randomization.
* 7. Capable of signing the informed consent form.

Exclusion Criteria:

* 1. New chronic heart failure patients, or patients receiving standard therapy on chronic heart failure for less than 3 months.
* 2. NYHA functional class I OR IV.
* 3. NT-proBNP < 600 pg/ml OR NT-proBNP>1700 pg/ml (by Roche assay Kit in central lab).
* 4. Patients with hypertrophic cardiomyopathy, rheumatic heart disease, constrictive pericarditis, significant valvular pathological change or congenital heart diseases, primary or secondary severe pulmonary artery hypertension.
* 5. Ischemic heart failure without recanalization or with recanalization in recent six months.
* 6. Acute MI in the last 3 months.
* 7. Unstable angina.
* 8. Patients with acute pulmonary edema or acute hemodynamic disorder.
* 9. Chronic heart failure patients with acute hemodynamic disorder or acute decompensation in the last 1 month (symptoms and signs suggest worsening chronic heart failure and may require intravenous drug therapy).
* 10. Patients with right heart failure caused by pulmonary disease.
* 11. Patients diagnosed with pericardial effusion (>50 ml) or pleural effusion(>200 ml), or evidenced by Echocardiogram.
* 12. Cardiac surgery or cerebrovascular accident within recent six months.
* 13. Preparing for heart transplantation or CRT, or has received CRT.
* 14. Serious ventricular arrhythmia (sustained ventricular tachycardia or frequent paroxysmal ventricular tachycardia).
* 15.Diagnosis of perinatal or chemotherapy-induced cardiomyopathy in last 12 months.
* 16. Serious hepatic or renal dysfunction (bilirubin 1.5 times above the normal upper limit, AST or ALT 2 times above the normal upper limit, serum creatinine>2.0mg/dL, HBV or HCV positive).
* 17. Serum potassium <3.2 mmol/L or >5.5 mmol/L.
* 18. Systolic blood pressure <90mmHg or >160mmHg.
* 19. Women of childbearing age who have a pregnancy plan within 2 years (women of childbearing age are defined as women who have a pregnancy physiology).
* 20. Pregnant or lactating women.
* 21. Patients who participated in any clinical trial in the recent three months.
* 22. Subject with a life expectancy less than 6 months as assessed by the investigator.
* 23. Serious nervous system diseases (Alzheimer's disease, advanced Parkinsonism),lower limb defects, or deaf-mute.
* 24. History of any malignancy or suffering from cancer, or biopsy proven pre-malignant condition (e.g., DICS or cervical atypia).
* 25. Evidence (physical examination, chest X-ray (CXR), ECHO or other tests) shows some active malignancy or adenoidal hypertrophy or neoplasm that has an effect on heart function or the endocrine system, e.g., pheochromocytoma or hyperthyroidism (Thyroid nodules with normal thyroid function do not need to be excluded).
* 26. As judged by the investigator that the subject cannot complete the study or adhere to the study requirements (due to the management reasons or others).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year
  Including deaths from cardiovascular and non-cardiovascular causes, Log-Rank test was used for comparison between groups, and Kaplan-Meier survival curves were plotted; COX proportional hazard model was used to estimate the HR and its 95% confidence interval.

SECONDARY OUTCOMES:
Mortality caused by cardiovascular events | 1 year
  Log-Rank test was used for comparison between groups, and Kaplan-Meier survival curves were plotted; COX proportional hazard model was used to estimate the HR and its 95% confidence interval.
All-cause mortality of female subjects | 1 year
  Log-Rank test was used for comparison between groups, and Kaplan-Meier survival curves were plotted; COX proportional hazard model was used to estimate the HR and its 95% confidence interval.
All-cause mortality of male subjects | 1 year
  Log-Rank test was used for comparison between groups, and Kaplan-Meier survival curves were plotted; COX proportional hazard model was used to estimate the HR and its 95% confidence interval.
Percentage of all-cause re-hospitalization | 1 year
  The Kaplan-Meier curve was used to describe the cumulative incidence rate of the first re-hospitalization, and the differences between the two groups were compared using Log-Rank.
Percentage of Participants with re-hospitalization caused by worsening heart failure | 1 year
  The Kaplan-Meier curve was used to describe the cumulative incidence rate of the first re-hospitalization, and the differences between the two groups were compared using Log-Rank.
Change of NT-proBNP level at the 25th week and 52th week | 1 year
  The paired t test or signed rank sum test was used to compare the changes before and after treatment in each group, and the comparison between groups was performed by analysis of variance or Wilcoxon rank sum test.
New York Heart Association (NYHA) functional classification | 1 year
  For the NYHA cardiac functional grading after administration, summarize the number and percentage of subjects by different study visit period, compare the efficacy differences among test groups and control groups. In addition, calculate the changes of NYHA cardiac functional grade from baseline of the subjects. The intragroup changes will be analyzed by signed-rank sum test, intergroup comparison will be conducted by Wilcoxon test.

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Ph.D,MD, Principal Investigator — Fuwai Hospital and Cardiovascular Institute, Chinese Academy of Medical Sciences
Locations (65):
- China (65):
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Navy General Hospital, Beijing, Beijing Municipality
  - Beijing Jingmei Group General Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital and Cardiovascular Institute, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Hospital of Chongqing Three Gorges Medical College, Chongqing, Chongqing Municipality
  - Chongqing Emergency Medical Center, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Sun Yai-sen Memorial hospital Sun Yai-sen University, Guangzhou, Guangdong
  - Guangdong Second Provincial Central Hospital, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - The First People's Hospital of Zunyi, Zunyi, Guizhou
  - Haikou People's Hospital, Haikou, Hainan
  - The Third People's Hospital of Hainan Province, Sanya, Hainan
  - HanDan Central Hospital, Handan, Hebei
  - First Hospital of Handan, Handan, Hebei
  - 980 Hospital of PLA Joint Logistics Support Force (Bethune International Peace Hospital), Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The Third Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First People's Hospital of Luoyang, Luoyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - The First People's Hospital of Xinxiang, Xinxiang, Henan
  - Pepole's hospital of Xinzheng, Xinzheng, Henan
  - Zhengzhou First People's Hospital, Zhengzhou, Henan
  - Luoyang center hospital, Zhengzhou, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Second Hospital. University of South China, Hengyang, Hunan
  - The First Affiliated Hospital of Baotou Medical College of Inner Mongolia University of Science & Technology, Baotou, Inner Mongolia
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiujiang Hospital Affiliated to Nanchang University, Jiujiang, Jiangxi
  - Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Jilin Academy of Traditional Chinese Medicine, Changchun, Jilin
  - Jilin University Sino-Japanese Friendship Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Central hospital of minhang District, Shanghai, Shanghai Municipality
  - The Sixth People's Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Oriental hospital, Shanghai, Shanghai Municipality
  - Shanghai Yangpu District Central Hospital, Shanghai, Shanghai Municipality
  - The Central Hospital of Putuo District, Shanghai, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi cardiovascular disease hospital, Taiyuan, Shanxi
  - Taiyuan City Central Hospital, Taiyuan, Shanxi
  - Pepole's hospital of DeYang city, Deyang, Sichuan
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Wuqing pepole's hospital, Tianjing, Tianjing
  - Fourth Affiliated Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - The Third People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Hospital of Kunming Medical College, Kunming, Yunnan
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Quzhou people's hospital, Quzhou, Zhejiang